CLINICAL TRIAL: NCT06099158
Title: Danish Pragmatic Randomized Trial to Evaluate the Effect of HeartLogic-Guided Management on Heart Failure Outcomes
Acronym: DANLOGIC-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, MP, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DANLOGIC-HF
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Pragmatic; Heart disease; ICD; CRT-D; Pacemaker; Registry; HeartLogic
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to treatment allocation. Active-arm participants will be unblinded at the time of first HeartLogic alert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HeartLogic-guided management (Experimental): HeartLogic alerts will be transmitted to the study team, which will subsequently contact the participant to assess any treatment needs. Treatment needs will be assessed according to current clinical practice guidelines.
  Interventions: Other: HeartLogic
- Standard care (No Intervention): The control group will receive usual HF care in the Danish health system.

INTERVENTIONS:
Other: HeartLogic — HeartLogic alerts will be managed according to a standardized alert management guide to ensure uniform reactions to HeartLogic alerts.
  Arms: HeartLogic-guided management

SUMMARY:
The purpose of the study is to assess the impact of HeartLogic-guided management on clinical outcomes among patients implanted with an eligible cardiac device.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, randomized controlled trial. Eligible patients in Denmark will be randomized 1:1 to either HeartLogic-guided management or usual care. During the trial, patients in the HeartLogic arm will be contacted by the study team in case of any HeartLogic alerts for evaluation and treatment decisions. There will be no mandatory in-person visits scheduled in the trial. HeartLogic alerts will be managed according to a prespecified management guide. Trial data besides device-related data will be retrieved from the Danish nationwide health registries including baseline information and endpoint data. The control group will receive usual HF care in the Danish health system without the involvement of the study team. The study will comply with the standards of the CONSORT statement and the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Implanted with a CRT-D or ICD device that has HeartLogic capability and ability to change HeartLogic enablement per randomization
2. Age ≥18 years
3. Compliant with remote monitoring and not listed in the LATITUDE™ remote monitoring system as "not monitored"

Exclusion Criteria:

There are no specific exclusion criteria for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of hospitalization for heart failure or all-cause death (first event) | 42 months

SECONDARY OUTCOMES:
Composite endpoint of hospitalization for heart failure or all-cause death (recurrent events) | 42 months
Hospitalization for heart failure (first event) | 42 months
All-cause hospitalization | 42 months
All-cause mortality | 42 months

OTHER OUTCOMES:
Hospitalizations for heart failure (recurrent events) | 42 months
Hierarchical composite of all-cause mortality, total number of heart failure hospitalizations, and total number of all-cause hospitalizations | 42 months
All-cause readmission within 30 days after hospitalization for heart failure | 42 months
Hospitalization for any cardiovascular disease | 42 months
Hospitalization for any cardio-respiratory disease | 42 months
Hospitalization for atrial fibrillation | 42 months
Atrial fibrillation burden | 42 months
Hospitalization for cardiac arrest | 42 months
Ventricular tachyarrhythmia leading to anti-tachycardia pacing and/or shock | 42 months
Cardiovascular mortality | 42 months
Incident heart failure (among participants without heart failure at baseline) | 42 months
Days alive and out of hospital | 42 months
Length of hospital stay | 42 months
Use of guideline-directed medical therapy for heart failure | 42 months
HeartLogic alert rate | 42 months
Average HeartLogic index | 42 months
Median HeartLogic alert length | 42 months
% time in HeartLogic alert | 42 months
Maximal observed HeartLogic index | 42 months
Time from HeartLogic alert to clinical event | 42 months
Individual HeartLogic sensor trends | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Study Chair — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.